CLINICAL TRIAL: NCT05185427
Title: Characterizing Error in Pulse Oximetry by Comparing Skin Pigmentation With Pulse Oximeter and Arterial Line Reading Deviations in Intensive Care Unit Pediatric Patients
Brief Title: Pulse Oximetry and Skin Pigmentation - Peds
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2021-30541
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Pulse Oximetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with pulse oximetry readings: The research team will take a reflectance measurement on the same location that the most recent pulse oximetry measurement was taken. In addition, a reflectance measurement will be taken bilaterally for the nailbed, dorsal and ventral side of the digits, dorsal and ventral side of the hand, dorsal and ventral side of the forearm, lower leg, foot, and either side for the ear. The most recent pulse oximetry and arterial oxygen saturation readings will be accessed through the electronic medical records, those readings are generally conducted simultaneously and will provide comparison. The duration anticipated for an individual participant's participation is 1 day.

SUMMARY:
The investigators' study aims to study how melanin index (mx) affects the deviation between SpO2 and SaO2, which becomes generally greater as hypoxia increases. The studies reviewed grouped individuals by race or have assigned individuals into groups like "dark", "intermediate", or "light" to describe pigmentation. Both of these methods are neither standardized nor objective, looking for race identifiers when it is more useful to be considering skin pigmentation identifiers. Skin pigmentation is a spectrum and it should be treated as such when trying to characterize relationships involving measurable factors such as melanin index.

The investigators will similarly measure the deviation between SpO2 and SaO2 however novel in that the investigators will quantitatively measure skin pigmentation via a light reflectance measurement device by Photovault.

DETAILED DESCRIPTION:
Pulse oximetry is an essential tool within healthcare due to its impressive ability to detect low oxygen levels even before hypoxia manifests in a patient. Despite being a powerful tool, pulse oximetry has limitations. It is well known that nail polish or jaundice can interfere with pulse oximetry readings. This knowledge influences clinical practice in that providers are aware of the inaccurately low saturation readings associated with nail polish and jaundice. Alarmingly, several studies have reported that pulse oximetry also fails to read as accurately for patients who have greater levels of skin pigmentation.

One theory reported by Bickler et al. (2005) and Fiener et al. (2007) suggests that pulse oximetry accuracy decreases as hypoxia increases, where this deviation is further amplified in the presence of greater levels of skin pigmentation. Bickler et al. (2005) reported statistically significant differences in pulse oximeter readings on three different pulse oximeters. They found a small bias existed at blood oxygen saturations above 80% and increased as desaturation increased. Specifically, this bias over-estimated blood oxygenation in Black patients where Bickler et al. reported a bias as much as 8% at very low oxygen saturation. A similar trend has been reported by others. Clinically, a staggering number of COVID-19 patients fall victim to "silent" or "apathetic" hypoxemia, exhibiting minimal symptoms of concern upon presentation, but rapidly experience multi-organ failure and in the most unfortunate circumstance, death, in less than 48 hours. If not concerned at the moment, emergency departments suggest patients self-monitor their oxygen saturation at home and return for further evaluation if they record an oxygenation reading below the COVID-19 protocol threshold. What would be a difference of a couple percentage points of observed oxygenation levels with a pulse oximeter in patients with more skin pigmentation determines admission, access to the required care, and risks a delay in the necessary oxygen supplementation of patients. One paper has even suggested that clinicians should accept 95% oxygen saturation for Black patients as opposed to a threshold of 92% SpO2 to ensure proper oxygenation. In January 2021, the World Health Organization included the use of pulse oximeters to assess and identify patients that would require hospitalization for COVID-19. However, in February 2021, the FDA cautioned against using pulse oximeter oxygen readings to diagnose or rule out COVID-19 patients, questioning its reliability in clinically significant circumstances shortly after the New England Journal of Medicine reported that Black patients suffered from occult hypoxemia nearly three times as much than White patients.

The investigators' study aims to study how melanin index (mx) affects the deviation between SpO2 and SaO2, which becomes generally greater as hypoxia increases. The studies reviewed grouped individuals by race or have assigned individuals into groups like "dark", "intermediate", or "light" to describe pigmentation. Both of these methods are neither standardized nor objective, looking for race identifiers when it is more useful to be considering skin pigmentation identifiers. Skin pigmentation is a spectrum and it should be treated as such when trying to characterize relationships involving measurable factors such as melanin index.

The investigators will similarly measure the deviation between SpO2 and SaO2 however novel in that the investigators will quantitatively measure skin pigmentation via a light reflectance measurement device by Photovault.

ELIGIBILITY:
Inclusion Criteria:

* Currently being cared for in the University of Minnesota Masonic Children's Hospital Intensive Care Unit (ICU)
* Already have an arterial line in place
* ICU staff state that it would be a good time to approach possible participants

Exclusion Criteria:

* If members of the research team are unable to access and measure with the Photovault the area that was measured via pulse oximetry by the care team
* Patients who do not have SpO2 or SaO2 measurements

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Intensive Care Unit (ICU) patients, potentially including COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Difference between pulse oximetry saturation (SpO2) and arterial line saturation (SaO2) | 1 day
  The reflective index will be measured in percent reflectance via the Photovault. The SpO2 is measured via pulse oximetry by the healthcare team as percent oxygen saturation. The SaO2 is measured via Arterial Blood Gas, which is also measured by the healthcare team. SaO2 is also reported in percent oxygen saturation. The difference between SpO2 and SaO2 as a factor of the reflective index will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth Fischer, MD, Principal Investigator — University of Minnesota Medical School Department of Internal Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No